CLINICAL TRIAL: NCT01790412
Title: Gestational Diabetes. The Rol of Exercise in the Prevention
Brief Title: Gestational Diabetes: the Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, Yaiza Cordero Rodríguez, Gestational Diabetes. The Role of Exercise in the Prevention, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Technical University of Madrid
Record Dates: First submitted 2013-02-05; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Pregnancy
Keywords: pregnancy, exercise, gestational diabetes
MeSH Terms: conditions — Motor Activity; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Experimental): Three sessions per week:
  Supervised exercise program
  Interventions: Behavioral: Exercise group
- Control (No Intervention): Sedentary pregnant women

INTERVENTIONS:
Behavioral: Exercise group — Combined two land aerobic sessions and one aquatic activities session
  Arms: Exercise group

SUMMARY:
To assess the effectiveness of an exercise program developed during pregnancy (land/aquatic activities) aerobic and muscular tonification, on control to the prevention to Gestational Diabetes. And to assess if excessive maternal weight gain is an influence in the diagnostic.

DETAILED DESCRIPTION:
A clinical, randomized controlled trial was used. 342 pregnant women without obstetric contraindications accepted informed consent for inclusion in the study. Finally, 257 were studied, 101 in intervention group (IG, n= 101) and 156 in control group (GC, n= 156). A physical exercise program three times per week during pregnancy was developed. The duration of session was 60 minutes and 50 minutes in land and water, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* At week 8-14
* Adherence 80% (minimum) until the end of pregnancy

Exclusion Criteria:

* Contraindications appointed by American College of Obstetricians & Gynecologists (ACOG)
* No adherence

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 257 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
prevention gestational diabetes | weeks 24-30
  Oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Maternal weight gain | weeks 40-42
  Maternal weight gain above guidelines recommendations by Institute of Medicine and National Research Council (IOM)

OTHER OUTCOMES:
Other pregnancy outcomes | After delivery
  macrosomia, type of delivery, birth weight

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Barakat, PhD, Study Director — Technical University of Madrid; Yaiza Cordero, PhD Student, Principal Investigator — Technical University of Madrid
Locations (1):
- Technical University of Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Cordero Y, Mottola MF, Vargas J, Blanco M, Barakat R. Exercise Is Associated with a Reduction in Gestational Diabetes Mellitus. Med Sci Sports Exerc. 2015 Jul;47(7):1328-33. doi: 10.1249/MSS.0000000000000547. PMID 25333246